CLINICAL TRIAL: NCT02694627
Title: Bandebereho Father Groups: a Randomized Control Trial to Assess the Impact of Maternal, Newborn and Child Health Group Education for New and Expecting Fathers
Brief Title: Bandebereho Father Groups Randomized Control Trial in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Promundo, United States (Other)
Collaborators: Rwanda Men's Resource Center (Rwamrec) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 137D
Record Dates: First submitted 2016-02-19; First posted 2016-02-29 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Gender Relations; Prenatal Care; Partner Communication; Contraception; Violence
Keywords: gender, caregiving, MNCH, violence, sexual and reproductive health, parenting
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): See intervention description
  Interventions: Behavioral: MenCare+/Bandebereho fathers'/couples' group education
- Control (No Intervention): Participants randomized into the control arm are surveyed at the same time points as intervention participants, but do not receive any intervention.

INTERVENTIONS:
Behavioral: MenCare+/Bandebereho fathers'/couples' group education — MenCare+/Bandebereho is a 3 year project to engage men in maternal, newborn and child health (MNCH) and in sexual and reproductive health in Rwanda. A core component of the project is fathers'/couples' group education. The target participants are first-time parents or parents of young children living in 16 rural and semi-urban sectors selected by the implementing partner in collaboration with local authorities. The MenCare+/Bandebereho fathers'/couples' group education engages men in 15 weekly sessions of group discussion, critical reflection and interactive activities led by a trained facilitator using a curriculum developed by RWAMREC and Promundo and approved by the Rwandan Ministry of Health, adapted from the Program P Manual. Men's partners participate in 6-8 sessions. The sessions focus on men's role in MNCH, family planning, sharing household responsibilities, intimate partner violence, conflict resolution, family budgeting, and gender equality.
  Other Names: Program P
  Arms: Intervention

SUMMARY:
This study seeks to assess the impact of the MenCare+/Bandebereho fathers'/couples' group education intervention on men's attitudes towards, and participation in, sexual and reproductive health, maternal, newborn and child health, and equitable and non-violent relationships with their children and partners.

DETAILED DESCRIPTION:
This study seeks to assess the impact of the MenCare+/Bandebereho fathers'/couples' group education intervention on men's attitudes towards, and participation in, sexual and reproductive health, maternal, newborn and child health, and equitable and non-violent relationships with their children and partners. The MenCare+/ Bandebereho program is a multi-component comprehensive intervention being implemented by the Rwanda Men's Resource Center (RWAMREC) and Promundo-US, in collaboration with the Rwanda Ministry of Health and local authorities in Karongi, Musanze, Nyaruguru and Rwamagana districts. The proposed study will evaluate one component of the program, a 15-session group education intervention targeting young fathers and mothers. The impact of the fathers' group education will be assessed through a randomized control trial design with an intervention arm of men and women participating in the father groups and a control arm of men and women who do not participate in the intervention. The study will collect quantitative and qualitative data over a period of approximately three years.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 21-35 years
* Living with a partner
* Expectant (or soon to be) father or father of young children under-5
* Living in an area with a group facilitator

Exclusion Criteria:

- Participated in previous cycles of the same intervention

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2400 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Gender division of caregiving/domestic tasks (from questionnaire: a) composite capturing frequency of the respondent doing household or caregiving tasks; b) composite capturing how tasks are shared between partners). | 4 months post intervention
Men's participation in family planning and maternal, newborn and child health (from questionnaire: a) men's presence at antenatal care visits; b) women's reports of receiving partner support during pregnancy; c) use of family planning). | 4 months post intervention
Gender-related attitudes (from questionnaire: a continuous scale variable, adapted from the validated Gender Equitable Men (GEM) scale). | 4 months post intervention
Women's experiences of intimate partner violence (from: questionnaire: a composite capturing exposure to a standard set of violent acts by a partner). | 4 months post intervention

SECONDARY OUTCOMES:
Use of violence/harsh punishment against children (from questionnaire: a composite capturing respondents' use of various harsh discipline acts in the past month, adapted from the UNICEF MICS study). | 4 months post intervention
Relationship quality measured (from questionnaire: a) frequency of quarreling and b) quality scale adapted from the Decision Making in Low-Income Couples). | 4 months post intervention
Couple communication (from questionnaire: a composite capturing frequency of communication across multiple topics). | 4 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kate E Doyle, MA, Principal Investigator — Promundo-US; Ruti G Levtov, PhD, Principal Investigator — Promundo-US; Gary Barker, PhD, Principal Investigator — Promundo-US; Shamsi Kazimbaya, MA, Principal Investigator — formerly at Rwanda Men's Resource Center, now at Jhpiego

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Levtov RG, Doyle K, Bingenheimer JB, Lahiri S, Kazimbaya S, Karamage E, Sayinzoga F, Mutoni M, Rubayita CH, Barker G. Improved Relationship Quality, Equitable Gender Attitudes, and Reduced Alcohol Abuse as Key Mechanisms to Reduce Intimate Partner Violence in the Bandebereho Couples' Randomized Trial in Rwanda. Prev Sci. 2022 Nov;23(8):1495-1506. doi: 10.1007/s11121-022-01445-6. Epub 2022 Oct 11. PMID 36219325
- [Derived] Doyle K, Levtov RG, Barker G, Bastian GG, Bingenheimer JB, Kazimbaya S, Nzabonimpa A, Pulerwitz J, Sayinzoga F, Sharma V, Shattuck D. Gender-transformative Bandebereho couples' intervention to promote male engagement in reproductive and maternal health and violence prevention in Rwanda: Findings from a randomized controlled trial. PLoS One. 2018 Apr 4;13(4):e0192756. doi: 10.1371/journal.pone.0192756. eCollection 2018. PMID 29617375